CLINICAL TRIAL: NCT02040454
Title: The Use of Intravascular Paclitaxel for the Treatment of Distal Radial Artery Arteriovenous Access Fistula Stenosis: A Randomized Study (PaciFIST-2)
Brief Title: Paclitaxel for the Treatment of Distal Radial Artery Arteriovenous Access Fistula Stenosis (PaciFIST-2)
Acronym: PaciFIST-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: required catheters not available
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-13-532
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Arteriovenous Access Fistula Stenosis
MeSH Terms: interventions — Paclitaxel; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy Plus Paclitaxel (Active Comparator): Standard Therapy - heparin, angioplasty, stent
  Paclitaxel - single intravascular dose up to 20 mg
  Interventions: Drug: Paclitaxel; Procedure: Standard Therapy
- Standard Therapy Alone (Sham Comparator): heparin, angioplasty, stent
  Interventions: Procedure: Standard Therapy

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Standard Therapy Plus Paclitaxel
Procedure: Standard Therapy

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the use of intravascular paclitaxel, in addition to standard therapy, for the treatment of arteriovenous dialysis access fistula stenosis.

A fistulogram will be performed in standard fashion. The diagnostic component will include evaluation of the inflow artery, arterial anastomosis and full length of the fistula vein or graft, plus venous return up to the heart. The location, vessel size, lesion diameter and percent stenosis for each lesion will be recorded. Enrollment and randomization will occur at this point.

All patients will then receive standard therapy for their stenosis. This will include intravenous heparin administered in a standard dose of 70 units/kg. Lesions that respond poorly to angioplasty (>30% residual stenosis after angioplasty treatment with 2 inflations) will be stented. Stent selection will be based on clinical setting. Initial stent treatment will utilize an uncovered nitinol stent. Treatment of in-stent restenosis will include initial balloon angioplasty, and use of a covered stent (Viabahn, GORE, or Fluency, Bard). Documentation of location and type of treatment for each lesion treated will be recorded.

Once standard treatment is completed, the operating surgeon will be informed of the results of randomization: treatment (paclitaxel) or control. For subjects assigned to treatment, the whole fistula vein outflow segment of the fistula will be treated with paclitaxel.

The full length of the radial artery from 1 cm of its origin to fistula anatomosis will be treated with paclitaxel. In addition the anastomosis and first 4 cm of the fistula vein will be treated. Paclitaxel solution treatment of each lesion encountered will be attempted until the 20 mg Paclitaxel dose limit is met. The volume administered will depend on the diameter and length of the vessels treated. Maximization of the length of vessel and lesions treated will be undertaken when there are more lesions than can be accommodated by the 12 mg, 10 ml dose available.

A 5 F sheath, 20 cm in length, will be used to administer the paclitaxel. This will be advanced from its distal position in the radial artery over the guidewire so that the tip of the sheath is in the proximal radial artery.

Prior to removal of the sheath, a final angiographic study of all areas treated is performed to document patency and lesion appearance. Any additional lesions identified with this study are then treated appropriately following standard technique.

For the control group, instead of paclitaxel administration, a sham treatment period of 10 minutes is allowed to elapse followed by the performance of the final completion angiogram. Any additional lesions identified with this study are then treated appropriately following standard technique.

All patients will follow the same follow up evaluation schedule

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient or guardian able to provide a signed informed consent
* Stenosis of the radial artery or initial 4 cm of the cephalic or basilic vein fistula with the anastomosis in the wrist greater than or equal to 50% treated satisfactorily (less than 20% residual stenosis) with balloon angioplasty alone or balloon angioplasty and stent placement
* Secondary fistulogram: the patient will have at least one prior fistulogram of the fistula to be treated.
* Either gender

Exclusion Criteria:

* Women who are pregnant or who are expected to or might become pregnant
* Women of child-bearing potential who do not use contraception
* Life expectancy less than 12 months
* Known allergy to paclitaxel
* Known allergy to contrast media not previously demonstrated to be controllable with premedication on a prior study using contrast
* Known allergy to the pre-medications (dexamethasone, famotidine, diphenhydramine)
* Pre-fistulogram thrombosis of the fistula
* Thrombectomy of the fistula within 14 days of the procedure
* Patient receiving chemotherapy
* Patients with an immunodeficiency disease or condition
* Documented hypercoagulable state
* WBC < 2000/mm3
* Platelet count less than 100,000/mm3
* Chronic hepatitis or jaundice
* Simultaneous enrollment in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Revascularization. | 6 months
  Target lesion revascularization (TLR) is defined as the need for subsequent clinically driven repeat angioplasty, stent placement or other intervention to correct the recurrence of a stenosis at the site treated within 6 months of the initial treatment.
Target Segment Revascularization. | 6 months
  Target segment revascularization (TSR) is defined as the need for secondary clinically driven repeat angioplasty, stent placement or other intervention to correct the recurrence of a stenosis in the radial artery or peri-anastomotic segment of cephalic or basilica vein treated with paclitaxel.

SECONDARY OUTCOMES:
Safety | 6 months
  The overall serious adverse event (SAE) rate will be determined as well as the rate for each individual type of adverse occurrence or event.
Binary Restenosis | 6 months
  The development of recurrent stenosis of the site treated with angioplasty or angioplasty and stent followed by the paclitaxel controlled infusion. The presence of a binary stenosis is defined as a 50% decrease of the vessel diameter measured on the fistulogram
Primary Patency: Fistula | 6 months
  The interval from treatment until access thrombosis or repeat intervention treatment to maintain fistula function, or the abandonment of the fistula.
Primary Assisted Patency: Fistula | 6 months
  The interval from treatment until access thrombosis, loss or abandonment
Secondary Patency: Fistula | 6 months
  The interval from treatment until access loss or abandonment, or surgical revision that replaces the segment of graft or fistula treated.
Primary Patency: Lesion | 6 months
  The interval from treatment until the lesion treated requires any type of re-treatment or occludes.
Primary Patency: Radial Artery Segment | 6 months
  The interval from treatment until the radial artery inflow segment treated requires any type of re-treatment or occludes.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Wengerter, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States